CLINICAL TRIAL: NCT05335499
Title: A Phase 2a, Randomized, Double-blind, Study of TAS5315 in Chronic Spontaneous Urticaria Patients With an Inadequate Response to H1-antihistamines
Brief Title: A Phase 2a Study of TAS5315 in Patients With Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10063040
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TAS5315 Dose 1 (Experimental)
  Interventions: Drug: TAS5315 Dose 1
- TAS5315 Dose 2 (Experimental)
  Interventions: Drug: TAS5315 Dose 2
- TAS5315 Dose 3 (Experimental)
  Interventions: Drug: TAS5315 Dose 3
- AS5315 Dose 4 (Experimental)
  Interventions: Drug: TAS5315 Dose 4
- TAS5315 Dose 5 (Experimental)
  Interventions: Drug: TAS5315 Dose 5
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS5315 Dose 1 — Treatment period: oral administration for 12 weeks, QD
  Arms: TAS5315 Dose 1
Drug: TAS5315 Dose 2 — Treatment period: oral administration for 12 weeks, QD
  Arms: TAS5315 Dose 2
Drug: TAS5315 Dose 3 — Treatment period: oral administration for 12 weeks, QD
  Arms: TAS5315 Dose 3
Drug: TAS5315 Dose 4 — Treatment period: oral administration for 12 weeks, QD
  Arms: AS5315 Dose 4
Drug: TAS5315 Dose 5 — Treatment period: oral administration for 12 weeks, QD
  Arms: TAS5315 Dose 5
Drug: Placebo — * Screening period: oral administration for 2 weeks, QD
  * Treatment period: oral administration for 12 weeks, QD
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAS5315 in chronic spontaneous urticaria patients with an inadequate response to H1-antihistamines

DETAILED DESCRIPTION:
The main purpose of this study is to assess the efficacy of TAS5315 in chronic spontaneous urticaria patients with an inadequate response to H1-antihistamines compared with placebo as measured by the change from baseline in weekly Urticaria Activity Score (UAS7) at week 12

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 18 to 75 years
* Diagnosis of chronic spontaneous urticaria (CSU)
* Presence of itch and hives for at least 6 consecutive weeks prior to screening in spite of use of non-sedating H1-antihistamines for CSU
* UAS7 score ≥ 16 and HSS7 score ≥ 8 during 7 days prior to study entry
* In-clinic UAS ≥ 4 on study entry
* Willing and able to complete and Participate Daily for the duration of the study

Key Exclusion Criteria

* Diseases other than CSU with symptoms of urticaria or angioedema, including urticarial vasculitis, erythema multiforme, mastocytosis, or hereditary or acquired angioedema
* Atopic dermatitis, psoriasis, ichthyosis, or other skin disease associated with chronic itching
* Bleeding diathesis
* Uncontrolled hypertension disease states
* Treatment with omalizumab or other humanized anti-human IgE monoclonal antibody therapies used to treat CSU within 4 months prior to screening
* Nonresponse to omalizumab or other humanized anti-human IgE monoclonal antibody therapies
* Have been treated with other Bruton's Tyrosine Kinase inhibitors
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in weekly Urticaria Activity Score (UAS7) at week 12 | Week 12
  The UAS7 is the sum of the HSS7 score (weekly Hives Severity Sore) and the ISS7 score (weekly Itch Severity Score). The range of the UAS7 score is 0 - 42.
  (Zuberbier et al. 1995; Zuberbier et al., 2014)

SECONDARY OUTCOMES:
Complete absence of hives and itch (UAS7=0) | Over time from week 1 to week 12
Disease control (UAS7<=6) | Over time from week 1 to week 12
Mean change from baseline in weekly Angioedema Activity Score (AAS7) | Over time from week 1 to week 12
  The AAS is a validated tool to assess occurrence of episodes of angioedema. The AAS7 is a weekly AAS score (AAS7). Minimum and maximum possible AAS7 scores are 0-105.
Mean change from baseline in Dermatology life quality index (DLQI) | Over time from week 1 to week 12
  DLQI is a 10-item dermatology-specific quality of life (QoL) measure. The range of the DLQI score is 0 - 30.
Mean change from baseline in Urticaria control test (UCT) | Over time from week 1 to week 12
  UCT is 4-item measure, which assesses symptoms, quality of life, treatment effectiveness. The range of the UCT score is 0 - 16.
Mean change from baseline in pharmacodynamics marker | Over time from week 1to week 12
  Pharmacodynamics marker are IgG, IgM, IgA, IgE, CRP and D-dimer.

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (12):
- Japan (12):
  - A site selected by Taiho Pharmaceutical Co., Ltd., Ehime
  - A site selected by Taiho Pharmaceutical Co., Ltd., Fukuoka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Gunma
  - A site selected by Taiho Pharmaceutical Co., Ltd., Hiroshima
  - A site selected by Taiho Pharmaceutical Co., Ltd., Ishikawa
  - A site selected by Taiho Pharmaceutical Co., Ltd., Kagawa
  - A site selected by Taiho Pharmaceutical Co., Ltd., Kumamoto
  - A site selected by Taiho Pharmaceutical Co., Ltd., Obihiro
  - A site selected by Taiho Pharmaceutical Co., Ltd., Osaka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Sapporo
  - A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo
  - A site selected by Taiho Pharmaceutical Co., Ltd., Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Taiho provides a platform for accepting researchers' requests for sharing anonymized, patient-level, analyzable datasets from articles published in peer-reviewed journals about the primary results from Taiho-sponsored interventional clinical trials in patients in which the medicine and the indication has received marketing approval from regulatory authorities in the United States, the European Union, and/or Japan on or after January 15, 2018.
Supporting Information: Study Protocol, SAP
Time Frame: https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html
Access Criteria: Access to the clinical trial data is contingent upon approval of a proposed study protocol by an independent review panel and the execution of a data-sharing agreement with the researcher.
URL: https://vivli.org/

REFERENCES:
- [Background] Zuberbier T, Chantraine-Hess S, Hartmann K, Czarnetzki BM. Pseudoallergen-free diet in the treatment of chronic urticaria. A prospective study. Acta Derm Venereol. 1995 Nov;75(6):484-7. doi: 10.2340/0001555575484487. PMID 8651031
- [Background] Zuberbier T, Aberer W, Asero R, Bindslev-Jensen C, Brzoza Z, Canonica GW, Church MK, Ensina LF, Gimenez-Arnau A, Godse K, Goncalo M, Grattan C, Hebert J, Hide M, Kaplan A, Kapp A, Abdul Latiff AH, Mathelier-Fusade P, Metz M, Nast A, Saini SS, Sanchez-Borges M, Schmid-Grendelmeier P, Simons FE, Staubach P, Sussman G, Toubi E, Vena GA, Wedi B, Zhu XJ, Maurer M; European Academy of Allergy and Clinical Immunology; Global Allergy and Asthma European Network; European Dermatology Forum; World Allergy Organization. The EAACI/GA(2) LEN/EDF/WAO Guideline for the definition, classification, diagnosis, and management of urticaria: the 2013 revision and update. Allergy. 2014 Jul;69(7):868-87. doi: 10.1111/all.12313. Epub 2014 Apr 30. PMID 24785199